CLINICAL TRIAL: NCT01020331
Title: Phase IIA Open Label Trial of Memantine in Combination With Riluzole (Customary Care) for the Treatment of ALS
Brief Title: Memantine Therapy in Amyotrophic Lateral Sclerosis
Acronym: TAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Phoenix Neurological Associates, LTD (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Todd Levine, MD, Phoenix Neurological Associates, LTD
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Memantine in ALS
Expanded Access: Available
Record Dates: First submitted 2009-11-20; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Memantine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ACTIVE (Experimental)
  Interventions: Drug: Memantine

INTERVENTIONS:
Drug: Memantine

SUMMARY:
Tau, a protein in the cerebrospinal fluid CSF is believed to be elevated in amyotrophic lateral sclerosis (ALS) patients. The investigators believe that Tau is truly a marker of increased neuronal death from any disease process. It is been shown that Memantine can inhibit and reverse the abnormal hyperphosphorylation of Tau and therefore the investigators are looking at the efficacy of Memantine at 10 mg twice a day (BID) to see if disease progression correlates with possible changes in Tau in ALS patients based on ALS Functional Rating Scale (ALSFRS) scores.

DETAILED DESCRIPTION:
We have been very interested in the role of developing a more active anti-excitotoxic cocktail for patients with ALS. As part of this interest we have been investigating potential markers for disease progression. One of our candidate markers has been the presence of elevated levels of TAU in the CSF of patients with ALS. While the presence of Tau was originally described as being used for adjunctive diagnostic testing in patients with Alzheimer's disease it has become clear that many neurodegenerative diseases possess elevated levels of Tau in the CSF. Therefore Tau is truly a marker of increased neuronal death from any disease process.

While levels of Tau have not been studied in depth in ALS, there was one report in 2003 which showed that 70% of ALS patients have elevated levels of Tau in their CSF (Sussmuth et al). We have also collected a series of 24 patients with clinically definite ALS and found that 22 of them had elevated levels of Tau at the time of diagnosis.

We have been intrigued by the findings that Memantine, an NMDA receptor antagonist, can inhibit and reverse the abnormal hyperphosphorylation of Tau which leads to sequestration of the normal Tau microtubules as well as microtubule associated protein 1 (MAP-1) and MAP-2. Further, Memantine has been shown to block the disassembly of microtubules which follows the hyperphosphorylation if Tau (Li et al., 2004).

We have submitted for presentation to the International Motor Neuron Disease meeting in 2005 the data on two anecdotal cases of patients with ALS. These two patients were diagnosed with ALS on clinical and electrophysiological data and they were found to have elevated levels of Tau in their CSF at the time of diagnosis. Both patients were treated with Riluzole, as standard therapy, and with Memantine 10 mg BID for 6 months. After 6 months their disease course was clearly very slow. A repeat analysis of their CSF showed that levels of Tau had returned to normal.

ELIGIBILITY:
Inclusion Criteria

1. Age 18-85
2. Male or Female
3. Clinically definite ALS by El Escorial criteria
4. Elevated levels of Tau in CSF

Exclusion Criteria:

1. Patients with FVC below 1.5 L or who require respiratory assistance
2. History of liver disease
3. Severe renal failure
4. History of intolerance to Riluzole or Memantine
5. Any other co morbid condition which would make completion of trial unlikely
6. If female, pregnant or breast-feeding; or, if of childbearing age, an unwillingness to use birth control.
7. Taking any trial medications. Non-trial medications are not cause for exclusion.
8. Unwillingness to provide consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-06; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Standardized assessment of ALS disease progression through the ALS Functional Rating Scale (ALSFRS) and compare the levels of Tau at baseline, 6 and 12 months | 18 months

SECONDARY OUTCOMES:
Change in muscle strength as measured by quantitative dynamometry (baseline vs 18 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Phoenix Neurological Associates, LTD, Phoenix, Arizona, United States